CLINICAL TRIAL: NCT01595841
Title: A Randomized Open Label Trial of Oral Sirolimus for Decrease of Stenosis in Arteriovenous Fistula in Hemo-dialysis Patients When Compared With Standard Therapy
Brief Title: Sirolimus Use in Angioplasty for Vascular Access Extension
Acronym: SAVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R-11-774; 17839 (Other: REB)
Record Dates: First submitted 2012-05-02; First posted 2012-05-10 (Estimated); Last update posted 2022-05-16 (Actual); Status verified 2022-04

CONDITIONS: End Stage Renal Disease; Venous Stenosis
Keywords: hemodialysis; stenosis; angioplasty; sirolimus
MeSH Terms: conditions — Kidney Failure, Chronic; Constriction, Pathologic | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sirolimus (Experimental): Participants will take sirolimus for 3 days prior to procedure and 30 days post procedure.
  Interventions: Drug: Sirolimus
- Not taking Sirolimus (No Intervention): Participants will not change the standard of care.

INTERVENTIONS:
Drug: Sirolimus — 3 mg po od loading dose for two days, then 2 mg po od for thirty days
  Other Names: rapamycin
  Arms: Sirolimus

SUMMARY:
Dialysis patients presenting for angioplasty intervention for graft failure will be randomized to receive either Sirolimus or not receive Sirolimus (standard of care) to assess the time from primary failure or angioplasty intervention to second or next angioplasty intervention or graft failure.

DETAILED DESCRIPTION:
This is a randomized control study to determine the feasibility of using sirolimus peri-angioplasty to compare the time from primary failure or angioplasty intervention to second or next angioplasty intervention or graft failure to a control group who would not have received Sirolimus

ELIGIBILITY:
Inclusion

1. hemodialysis patients referred for angioplasty for hemodialysis access stenosis through either access flow or clinical monitoring in either an AVF or AVG
2. > 18 years of age.
3. Total white blood cell count > 3 x 109 /L and platelet count > 100.0 x 103/uL
4. Fasting triglycerides < 4.0 mmol/L, fasting cholesterol < 7.8 mmol/L while on optimal lipid lowering therapy.

Exclusion Criteria:

1. A woman who is pregnant or breastfeeding
2. Active malignancy
3. Concomitant treatment with immunosuppressant medications
4. Active infection or treated for infection within the last 30 days
5. Pre-existing interstitial lung disease
6. Thrombocytopenia with platelets less than 100 109/L
7. Previous renal or other solid organ transplant
8. Preexisting liver failure
9. Life expectancy less than 6 months
10. Planned major surgery or major surgery within the last 6 months
11. History of malignancy within the previous 5 years (with the exception of adequately treated basal cell or squamous cell carcinoma of the skin).
12. Known history of any coronary intervention within the 6 months prior to current screening
13. Prior or current use of Sirolimus or any of its derivatives within 3 months prior to angioplasty
14. Active gastrointestinal disorder that may interfere with drug absorption
15. Known to be HIV positive or known active hepatitis B or C infection
16. Treatment with voriconazole, terfenadine, cisapride, astemizole, pimozide, or ketoconazole (known to interact with Sirolimus) that is not discontinued before starting Sirolimus treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-12; Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Comparison of the sirolimus group to the control group from time of assisted primary and secondary patency rates to access abandonment | 12 months
  Comparison of the sirolimus group to the control group from time of assisted primary and secondary patency rates to access abandonment

SECONDARY OUTCOMES:
Secondary End point | 12 months
  Secondary end points will be improvement in vascular access flow rates as measured by either online conductivity dialysance or ultrasound dilution techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Jevnikar, MSc MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol